CLINICAL TRIAL: NCT07051252
Title: A Phase 1b, Open-Label Study of HBS-201 (Pitolisant Delayed-release) in Adult Participants With Narcolepsy
Brief Title: A Study of HBS-201 (Pitolisant Delayed-release)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Harmony Biosciences Management, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HBS-101DR-CL-101
Record Dates: First submitted 2025-06-30; First posted 2025-07-04 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Narcolepsy
Keywords: Narcolepsy; Pitolisant hydrochloride; Pitolisant delayed-release
MeSH Terms: conditions — Narcolepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- HBS-201 (Experimental): Participants will take HBS-201 orally once daily in the morning upon wakening, beginning the morning of Day 1 and continuing through Day 14.
  Interventions: Drug: HBS-201

INTERVENTIONS:
Drug: HBS-201 — On Days 1-7, participants will take HBS-201 17.8 mg per day (one 17.8 mg tablet) and on Days 8-14, participants will take HBS-201 35.6 mg per day (two 17.8 mg tablets).
  Other Names: pitolisant delayed-release (DR); pitolisant hydrochloride

SUMMARY:
The purpose of this study is to assess the tolerability of HBS-201 when starting at a therapeutic dose in adult participants with narcolepsy.

DETAILED DESCRIPTION:
This is a Phase 1b, open-label, multicenter study to assess the tolerability of HBS-201 when starting at a therapeutic dose in adult participants with narcolepsy. Therapeutic dose range is defined as 17.8 milligram (mg) to 35.6 mg based on the FDA-approved prescribing information for WAKIX.

The study will consist of an up to 30-day Screening/Baseline Period, a 2-week Open-Label Period, and a 30-day Safety Follow-up Period.

ELIGIBILITY:
Inclusion Criteria:

1. Has a current documented diagnosis of narcolepsy type 1 or narcolepsy type 2 per International Classification of Sleep Disorders, 3rd Edition (ICSD-3) criteria.

Exclusion Criteria:

1. Has hypersomnolence due to another medical disorder.
2. Is currently taking or has taken WAKIX (pitolisant).
3. Has participated in an interventional research study involving another investigational medication, device, or behavioral treatment within 30 days or within 5 half-lives of the investigational medication prior to Screening.
4. Based on the judgment of the Investigator, is unsuitable for the study for any reason, including but not limited to unstable or uncontrolled medical conditions (including psychiatric and neurological conditions) or a medical condition that might interfere with the conduct of the study, confound interpretation of study results, pose a health risk to the participant, or compromise the integrity of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2025-05-21 (Actual); Primary Completion 2025-10-13 (Actual); Study Completion 2025-10-13 (Actual)

PRIMARY OUTCOMES:
Percentage of participants who discontinue treatment due to a treatment-emergent adverse event (TEAE) related to study drug | From administration of the first dose of study drug (Day 1) through 30 days after the final dose of study drug, approximately 44 days
  A TEAE is any adverse event (AE) reported after the first dose of study drug, or any worsening of a pre-existing condition reported after first dose of study drug.
Frequency, severity, and seriousness of TEAEs | From administration of the first dose of study drug (Day 1) through 30 days after the final dose of study drug, approximately 44 days
  A TEAE is any adverse event (AE) reported after the first dose of study drug, or any worsening of a pre-existing condition reported after first dose of study drug.

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - Harmony Site 9, San Ramon, California
  - Harmony Site 14, Brandon, Florida
  - Harmony Site 4, Miami, Florida
  - Harmony Site 8, Atlanta, Georgia
  - Harmony Site 13, Newton, Massachusetts
  - Harmony Site 11, Troy, Michigan
  - Harmony Site 10, Denver, North Carolina
  - Harmony Site 2, Huntersville, North Carolina
  - Harmony Site 6, Canton, Ohio
  - Harmony Site 1, Cincinnati, Ohio
  - Harmony Site 15, Wyomissing, Pennsylvania
  - Harmony Site 5, Columbia, South Carolina
  - Harmony Site 12, North Charleston, South Carolina
  - Harmony Site 3, Austin, Texas
  - Harmony Site 7, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: No